CLINICAL TRIAL: NCT06356350
Title: Effects of Exercise Programs on Gait in Children With Juvenile Idiopathic Arthritis
Brief Title: Exercise Programs on Gait in Children JIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gokce Leblebici, Principal investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IUC_jia_gait
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Juvenile Idiopathic Arthritis; Gait, Frontal
Keywords: juvenile idiopathic arthritis; gait; exercise; physiotherapy
MeSH Terms: conditions — Arthritis, Juvenile; Gait Disorders, Neurologic; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core based exercise group (Active Comparator): This group will be undergone core based exercises program
  Interventions: Other: Core based exercises
- Neuromuscular exercises group (Active Comparator): This group will be undergone conventional neuromuscular exercises program
  Interventions: Other: Conventional neuromuscular exercises

INTERVENTIONS:
Other: Conventional neuromuscular exercises — Conventional neuromuscular exercises represent a contemporary physiotherapeutic approach. These exercises aim to improve neuromuscular control, strength, and endurance in various muscles surrounding the included joint, contributing to the correction and maintenance of proper posture.
  Arms: Neuromuscular exercises group
Other: Core based exercises — Core based exercises increase overall mobility, relieve pain, improve posture, and support spinal alignment. Especially important for children who are still growing is to slow or stop the progression of deformities because of the asymmetrical loading pattern.
  Arms: Core based exercise group

SUMMARY:
Juvenile Idiopathic Arthritis (JIA) is one of the common chronic diseases in childhood. Problems such as weakness or pain may occur in JIA, especially in the joints and the muscles around the trunk. These conditions may lead to abnormal displacement of the center of gravity, deterioration of biomechanics, and muscle imbalance in children with JIA. All these situations can lead to postural imbalance and asymmetrical loading pattern, which we often encounter in children with JIA. Current studies describing various exercise methods effective on postural alignment. However, no study was found in the literature that searching the effects of these exercise methods on gait parameters in children JIA.

DETAILED DESCRIPTION:
Juvenile Idiopathic Arthritis (JIA) is one of the common chronic diseases in childhood. Problems such as weakness or pain may occur in JIA, especially in the joints and the muscles around the trunk. These conditions may lead to abnormal displacement of the center of gravity, deterioration of biomechanics, and muscle imbalance in children with JIA. These conditions may lead to abnormal displacement of the center of gravity, deterioration of biomechanics, and muscle imbalance in children with JIA. All these situations can lead to postural imbalance and asymmetrical loading pattern, which we often encounter in children with JIA. Current studies describing various exercise methods effective on postural alignment. However, no study was found in the literature that searching the effects of these exercise methods on gait parameters in children JIA. Therefore, this study aimed to investigate the effects of two different exercise programs (core based exercise program against neuromuscular training) on gait parameters in children JIA.

In this study, the participants will be evaluated and then they will be divided into two groups randomly. The first group will be administered as a core based exercise program group and the second one will be undergone as a neuromuscular training group. After the interventions, they will be re-evaluted by the physiotherapist and the outcomes will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Having a diagnosis of oligoarticular JIA
* Being between the age of 8 and 16
* Having included knee joint.

Exclusion Criteria:

* Having an additional neurological or orthopedic diagnosis other than JIA Affecting treatment results,
* Having had any surgery on the spine or the extremity joints
* Being at a level that will not understand the questions asked.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
Maximum Loading | immediately after intervention
  It will be obtained using the FreeMed baropodometry platform (the FreeStep v. 1.0. 3 88 software, Sensor Medica, Guidonia Montecelio, Roma, Italy). The unit of the outcome is per cent.
Center of mass displacement | immediately after intervention
  It will be obtained using the FreeMed baropodometry platform (the FreeStep v. 1.0. 3 88 software, Sensor Medica, Guidonia Montecelio, Roma, Italy). The unit of the outcome is milimeter.
Walking speed | immediately after intervention
  It will be obtained using the FreeMed baropodometry platform (the FreeStep v. 1.0. 3 88 software, Sensor Medica, Guidonia Montecelio, Roma, Italy). The unit of the outcome ia meter/second.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ombrello MJ, Arthur VL, Remmers EF, Hinks A, Tachmazidou I, Grom AA, Foell D, Martini A, Gattorno M, Ozen S, Prahalad S, Zeft AS, Bohnsack JF, Ilowite NT, Mellins ED, Russo R, Len C, Hilario MO, Oliveira S, Yeung RS, Rosenberg AM, Wedderburn LR, Anton J, Haas JP, Rosen-Wolff A, Minden K, Tenbrock K, Demirkaya E, Cobb J, Baskin E, Signa S, Shuldiner E, Duerr RH, Achkar JP, Kamboh MI, Kaufman KM, Kottyan LC, Pinto D, Scherer SW, Alarcon-Riquelme ME, Docampo E, Estivill X, Gul A; British Society of Pediatric and Adolescent Rheumatology (BSPAR) Study Group, Inception Cohort of Newly Diagnosed Patients with Juvenile Idiopathic Arthritis (ICON-JIA) Study Group, Childhood Arthritis Prospective Study (CAPS) Group, Randomized Placebo Phase Study of Rilonacept in sJIA (RAPPORT) Investigators, Sparks-Childhood Arthritis Response to Medication Study (CHARMS) Group, Biologically Based Outcome Predictors in JIA (BBOP) Group; Langefeld CD, Thompson S, Zeggini E, Kastner DL, Woo P, Thomson W. Genetic architecture distinguishes systemic juvenile idiopathic arthritis from other forms of juvenile idiopathic arthritis: clinical and therapeutic implications. Ann Rheum Dis. 2017 May;76(5):906-913. doi: 10.1136/annrheumdis-2016-210324. Epub 2016 Dec 7. PMID 27927641
- [Background] Tokuda K, Anan M, Takahashi M, Sawada T, Tanimoto K, Kito N, Shinkoda K. Biomechanical mechanism of lateral trunk lean gait for knee osteoarthritis patients. J Biomech. 2018 Jan 3;66:10-17. doi: 10.1016/j.jbiomech.2017.10.016. Epub 2017 Nov 4. PMID 29150344
- [Background] Ringold S, Wallace CA, Rivara FP. Health-related quality of life, physical function, fatigue, and disease activity in children with established polyarticular juvenile idiopathic arthritis. J Rheumatol. 2009 Jun;36(6):1330-6. doi: 10.3899/jrheum.081028. Epub 2009 May 1. PMID 19411394
- [Background] KISA, E. P., & OTMAN, A. S. (2020). Skolyoz odaklı egzersizler-yedi büyük okulun kapsamlı incelemesi. Süleyman Demirel Üniversitesi Sağlık Bilimleri Dergisi, 11(2), 255-259.
- [Background] Horng J, Liu XC, Thometz J, Tassone C, Duey-Holtz A. Evaluation of plantar pressures and center of pressure trajectories in Adolescent Idiopathic Scoliosis. Stud Health Technol Inform. 2021 Jun 28;280:131-135. doi: 10.3233/SHTI210451. PMID 34190074
- [Background] Gao CC, Chern JS, Chang CJ, Lai PL, Lung CW. Center of pressure progression patterns during level walking in adolescents with idiopathic scoliosis. PLoS One. 2019 Apr 22;14(4):e0212161. doi: 10.1371/journal.pone.0212161. eCollection 2019. PMID 31009471
- [Background] Zhu F, Hong Q, Guo X, Wang D, Chen J, Zhu Q, Zhang C, Chen W, Zhang M. A comparison of foot posture and walking performance in patients with mild, moderate, and severe adolescent idiopathic scoliosis. PLoS One. 2021 May 17;16(5):e0251592. doi: 10.1371/journal.pone.0251592. eCollection 2021. PMID 33999943